CLINICAL TRIAL: NCT06223672
Title: Essential Fats For Enhancing Cognitive Thinking (EFFECT) Study: Dietary Fat Quality and Cognitive Impairment
Brief Title: Essential Fats For Enhancing Cognitive Thinking (EFFECT) Study
Acronym: EFFECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); The California Walnut Commission (Unknown)
Responsible Party: Principal Investigator, Martha Belury, Professor and Chair, Food Science and Technology, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023H0111
Record Dates: First submitted 2023-10-09; First posted 2024-01-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Decline; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Walnuts (Experimental): consumption of walnuts every day
  Interventions: Other: Walnuts
- White chocolate-style bar (Experimental): consumption of a white chocolate-style bar every day
  Interventions: Other: Simply White Diary-free chocolate bar

INTERVENTIONS:
Other: Walnuts — 56g of walnuts consumed each day for 7 days
  Arms: Walnuts
Other: Simply White Diary-free chocolate bar — 68g of the white chocolate style-bar each day for 7 days
  Arms: White chocolate-style bar

SUMMARY:
The proposed research is a randomized crossover trial designed to assess changes in postprandial cognitive function and the gut-brain axis in adults with subjective cognitive complaints who consume 1 study snack per day for 1 week.

DETAILED DESCRIPTION:
Study objective including

1. To measure the impact of dietary fats on postprandial cognitive function in adults who report subjective cognitive complaints.
2. To assess the effect of dietary fat consumption on the gut-brain axis in relationship to cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Subjective cognitive impairment
* BMI ≥30 kg/m2
* HbA1C <6.5%

Exclusion Criteria:

* Diagnosis og cognitive impairment or dementia
* Montreal Cognitive Assessment (MoCA) score of <26
* Current or previous diagnosis of Diabetes or use of diabetes medications
* Current diagnosis of or current treatment of cancer other than non-melanoma skin cancer
* Gastrointestinal diseases or disorders (including pancreatic and gastric bypass surgery) where consumption of the study foods would be contraindication or where the disease or disorder could negatively affect nutrient absorption and/or would prevent participants from tolerating the study foods
* Hyperthyroidism diagnosis
* Food Allergy or intolerances
* Any dietary restriction where consumption of the study foods, study meals/snack or meal challenge or any ingredient would be contraindicated
* Use of some oil supplements in the past 4 weeks prior to enrolling
* Pregnancy and lactation
* Inability to access veins for venipuncture
* Antibiotic use in the past month
* Psychostimulant or nootropic medication use
* Current use of supplements or medications for weight loss or following a weight loss program
* Severe or uncontrolled autoimmune diseases
* Current or previous diagnosis of severe kidney failure, liver cirrhosis and some pulmonary diseases
* Heart disease events (including stroke or heart attack) within last 3 months prior to enrollment
* Alcohol or drug abuse

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function measured using the National Institutes of Health Toolbox for the Assessment of Neurological and Behavioral Function Cognitive Battery (NIHTB-CB) | Week 0 and Week 5
  To determine the impact of consuming the study dietary fats as part of a high fat meal on postprandial cognitive function

SECONDARY OUTCOMES:
Change in Cognitive function measured using the National Institutes of Health Toolbox for the Assessment of Neurological and Behavioral Function Cognitive Battery (NIHTB-CB) | Week 0, Week 1, Week 5 and Week 6
  To assess changes in cognitive function after consuming 1 serving of the dietary fats every day for 1 week
Changes in fecal Microbiota diversity | Week 0, Week 1, Week 5 and Week 6
  To assess changes in microbiota diversity of fecal samples after consuming 1 serving of the dietary fats every day for 1 week

OTHER OUTCOMES:
Changes in postprandial energy metabolism | Week 0 and Week 5
  To evaluate the effect of dietary fats on postprandial indirect calorimetry (kilocalories)
Changes in postprandial respiratory quotient | Week 0 and Week 5
  To evaluate the effect of dietary fats on postprandial respiratory quotient to identify what fuels (carbohydrate protein or fat) are utilized
Changes in postprandial lipids | Week 0 and Week 5
  To evaluate the effect of dietary fats on postprandial lipid panel including total cholesterol, HDL-Cholesterol, LDL-Cholesterol, Triglycerides (mg/dL)
Changes in postprandial Tumor necrosis factor levels | Week 0 and Week 5
  To evaluate the effect of dietary fats on postprandial blood Tumor necrosis factor alpha (TNF), a marker of inflammation
Changes in postprandial IL-6 | Week 0 and Week 5
  To evaluate the effect of dietary fats on postprandial blood IL-6 a marker of inflammation
Changes in postprandial C-Reactive Protein | Week 0 and Week 5
  To evaluate the effect of dietary fats on postprandial blood C-reactive protein, a marker of inflammation
Changes in postprandial Soluble intercellular adhesion molecule-1 | Week 0 and Week 5
  To evaluate the effect of dietary fats on postprandial blood Soluble intercellular adhesion molecule-1, a marker of inflammation
Changes in cardiolipin species | Week 0, Week 1, Week 5 and Week 6
  To determine the impact of dietary fat on peripheral blood mononuclear cell cardiolipin species measured using electrospray ionization-mass spectrometry coupled to high-performance liquid chromatography
Changes in postprandial glucose levels | Week 0 and Week 5
  To determine the impact of dietary fat on postprandial blood glucose levels
Changes in postprandial insulin levels | Week 0 and Week 5
  To determine the impact of dietary fat on postprandial blood insulin levels
Changes in postprandial cortisol levels | Week 0 and Week 5
  To determine the impact of dietary fat on postprandial salivary cortisol levels

CONTACTS AND LOCATIONS:
Overall Officials: Martha Belury, PhD, RDN, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Zarich S, Cole RM, Fairchild K, Spakowicz D, Sparagna G, Madison A, Ni A, Belury MA. Effects of Walnuts on Postprandial Cognitive Function in Adults With Subjective Cognitive Impairment: Protocol for a Randomized Crossover Trial. JMIR Res Protoc. 2025 Dec 19;14:e82032. doi: 10.2196/82032. PMID 41418290